CLINICAL TRIAL: NCT06921824
Title: Investigating the Effect of Glucagon on Cognitive Function and Cerebral Glucose Metabolism in Humans: A Pilot Study
Brief Title: Investigating the Acute Effects of Increasing Glucagon Exposure in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Principal Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GluCoMet_stepwise glucagon
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glucose Metabolism; Glucagon
MeSH Terms: interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucagon Infusion (Experimental)
  Interventions: Other: Glucagon

INTERVENTIONS:
Other: Glucagon — A three-hour intravenous infusion with glucagon with increasing infusion rate (from 0,01 ng/kg/min up to 50 ng/kg/min)

SUMMARY:
In this study the investigators will investigate the acute effects of increasing glucagon exposure on metabolic parameters in healthy participants.

Participants will participate in one study day. After initial baseline blood samples, a three-hour intravenous infusion with glucagon will be initiated. The infusion rate will be increased every 30 minutes.

DETAILED DESCRIPTION:
Ten participants with normal health will be included, and each participant will participate in one study day.

Participants will arrive after an overnight fast and will be placed in a hospital bed in a semi-recumbent position. In each antecubital vein an intravenous catheter will be placed; one for administration of glucagon and one for blood sampling.

Two baseline blood samples will be drawn before the glucagon infusion is started. The glucagon infusion rate will be increased every 30 minutes (infusion rates are 0,01 ng/kg/min, 0,1 ng/kg/min, 0,5 ng/kg/min, 1,0 ng/kg/min, 10 ng/kg/min and 50 ng/kg/min).

Blood samples for the analysis of plasma glucagon, glucose, insulin, C-peptide etc. will be drawn every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the participant information and signing the consent form
* Between 25 and 70 years of age at the time of screening
* Body mass index (BMI) ≤ 25 kg/m2 at the time of screening

Exclusion Criteria:

* Enrolment in other research projects that might interfere with the study
* Diabetes diagnosis (type 1 and 2)
* Pregnancy or breastfeeding
* Use of medications which, in the opinion of the investigator, may jeopardise participant's safety or compliance with the protocol
* Impaired liver function defined as either alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) ≥ 2 times normal values
* Kidney disease defined as serum creatinine levels ≥ 126 μmol/L for male and ≥ 111 μmol/L for female
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range 90-150 mmHg for systolic and 50-100 mmHg for diastolic
* Active or recent malignant disease
* Current or history of severe alcohol use or drug/chemical abuse as per investigator's judgement
* Any chronic disorders or severe diseases which, in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Glucagon infusion rate that increases plasma glucose | 0-180 minutes
  Glucagon infusion rate at which plasma glucose levels are significantly increased compared to baseline

SECONDARY OUTCOMES:
Glucagon infusion rate that increases plasma cAMP | 0-180 minutes
  Glucagon infusion rate at which plasma cAMP levels are significantly increased compared to baseline
Glucagon infusion rate that decreases plasma amino acids | 0-180 minutes
  Glucagon infusion rate at which plasma amino acid levels are significantly decreased compared to baseline
Glucagon infusion rate that affects plasma triglycerides | 0-180 minutes
  Glucagon infusion rate at which plasma triglycerides are significantly changed compared to baseline
Glucagon infusion rate that affects plasma nonesterified fatty acids | 0-180 minutes
  Glucagon infusion rate at which plasma nonesterified fatty acids are significantly changed compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai J Wewer Albrecthsen, MD PhD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
Locations (1):
- Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark, Copenhagen, Denmark